CLINICAL TRIAL: NCT03544879
Title: Yoga to Prevent Mobility Limitations in Older Adults: A Pilot Randomized Controlled Trial
Brief Title: Yoga to Prevent Mobility Limitations in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Erik Groessl, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130472
Record Dates: First submitted 2018-05-18; First posted 2018-06-04 (Actual); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Aging; Mobility Limitation; Sedentary Lifestyle
MeSH Terms: conditions — Mobility Limitation; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): The yoga intervention consisted of 2x weekly 60-minute sessions for 10 weeks. Yoga consists of postures, breathing exercises, movement, and meditation/concentration..
  Interventions: Behavioral: Yoga Intervention
- Health Education (Active Comparator): The health education comparison intervention consisted of once weekly, 90-minute health information workshops conducted in group format. Sessions generally consisted of a 60-minute lecture followed by 30 minutes of questions and discussion.
  Interventions: Behavioral: Healthy Aging Education

INTERVENTIONS:
Behavioral: Yoga Intervention — The 60-minute yoga sessions began with a brief breathing practice led by the instructor. The yoga instructor then led students through yoga poses at a gentle pace using chairs as props as needed. The pace of the class increased slowly over time as students became more familiar and more capable with the poses. Meditation and breathing was followed by chair poses (15-20 minutes), standing poses (10-15 minutes), floor poses (15 minutes), and lastly a supine resting pose (Savasana; 10 minutes). In the Silver Age Yoga method at that time, there were 73 available postures overall including: 35 Chair Postures, 18 Standing Postures, 20 Floor Postures, with a typical class covering 20-25 poses.
  Arms: Yoga
Behavioral: Healthy Aging Education — The health education comparison intervention consisted of once weekly, 90-minute health information workshops conducted in group format. The 90-minute sessions generally consisted of a 60-minute lecture followed by 30 minutes of questions and discussion. The lecture titles for Weeks 1-10 were as follows: Introduction/ Exploring Communication, The Science of Successful Aging, Acupuncture 101: How it Works & What it is Good for, Quality of Life/Quality of Well Being, Fighting Cancer With Your Fork, Forgiveness via Shakespeare's: A Winter's Tale, Better Eyesight in Minutes a Day, Brain Fitness, The Importance of Organic Foods/ Organic Gardening, How Dementia Can Be Modified. Lectures were provided by a mix of credentialed experts (physicians/psychologists, etc) and other clinicians. Instructors were asked not to talk about yoga or medication in their lectures. Content was not otherwise closely monitored.
  Arms: Health Education

SUMMARY:
The loss of mobility during aging impacts independence and leads to further disability, morbidity, and reduced life expectancy. The study objective was to examine the feasibility and safety of conducting a randomized controlled trial of yoga for older adults at risk for mobility limitations. The investigators hypothesized that sedentary older adults could be recruited for the study, would attend either yoga or a health education control, would complete assessments, and that the interventions could be safely delivered.

ELIGIBILITY:
Inclusion Criteria:

* age 60-89 years
* self-reported sedentary lifestyle (not exercising in the past 3 months; included walking at a brisk pace or regular walking for exercise purposes)
* SPPB summary score > 3 and ≤ 8
* willingness attend either yoga or health education for 10 weeks
* willing to complete two assessments
* residence in San Diego metropolitan area
* provided a physician-signed health clearance form.

Exclusion Criteria:

* practiced yoga > 2x in the last year
* life expectancy < 12 months.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2014-05-02 (Actual); Study Completion 2014-06-30 (Actual)

IPD SHARING:
Plan to Share IPD: No
Data is still being analyzed.

REFERENCES:
- [Derived] Groessl EJ, Maiya M, Schmalzl L, Wing D, Jeste DV. Yoga to prevent mobility limitations in older adults: feasibility of a randomized controlled trial. BMC Geriatr. 2018 Dec 12;18(1):306. doi: 10.1186/s12877-018-0988-8. PMID 30541474

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Education: The health education comparison intervention consisted of once weekly, 90-minute health information workshops conducted in group format. Sessions generally consisted of a 60-minute lecture followed by 30 minutes of questions and discussion.
  The lecture titles for Weeks 1-10 were as follows: Introduction/ Exploring Communication, The Science of Successful Aging, Acupuncture 101: How it Works & What it is Good for, Quality of Life/Quality of Well Being, Fighting Cancer With Your Fork, Forgiveness via Shakespeare's: A Winter's Tale, Better Eyesight in Minutes a Day, Brain Fitness, The Importance of Organic Foods/ Organic Gardening, How Dementia Can Be Modified. Lectures were provided by a mix of credentialed ex
Period: Overall Study
Arm/Group | Yoga | Health Education
Started | 22 | 24
Completed Follow-up Physical Assessment | 20 | 21
Completed (refers to completing follow-up self-report questionnaires) | 22 | 23
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga | Health Education | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (8.3) | 76.0 (7.8) | 73.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 7 | 11 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 0 | 1 | 1
  White | 18 | 20 | 38
  Native American | 1 | 0 | 1
  Asian/Pacific Islander | 0 | 1 | 1
  Hispanic | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery (SPPB) measures time to walk four meters; time to five chair stands; and balance, with higher scores being associated with decreased disability and mortality. These 3 components are rated on a scale from 0-4 and they are summed to provide a total SPPB score ranging from 0-12.
Time Frame: Change in SPPB from baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Health Education
Number analyzed (Participants) | 20 | 21
units on a scale | 1.55 (1.67) | 1.18 (1.33)

2. Secondary Outcome: Step Up and Over (SUO)
Description: The Step Up and Over (SUO) test measures gait quality as it may influence negotiating curbs, climbing or descending stairs, and predicting fall risk. The lift index quantifies the maximum lifting force exerted by the leading leg expressed as a percentage of the individual's weight as measured by the force plate, with scores closer to 100% demonstrating greater force.
Time Frame: Change from baseline to 10 weeks
Population: 2 participants in each group completed written self-report measures but not physical assessments at 10 weeks (follow-up).
Measure: Mean (Standard Deviation); unit: percent of weight
Arm/Group | Health Education | Yoga
Number analyzed (Participants) | 21 | 20
percent of weight | -0.65 (9.0) | 8.7 (26.3)

3. Secondary Outcome: Rhythmic Weight Shift (RWS)
Description: Rhythmic Weight Shift (RWS) measures participant ability to rhythmically move between two targets at different speeds. The On-Axis Velocity is the speed of the COG displacement in degrees per second during on-axis movement between the test target(s), with greater velocity indicating faster movement through the region of stability
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | Health Education | Yoga
Number analyzed (Participants) | 21 | 20
degrees per second | 0.07 (1.14) | -0.15 (0.83)

4. Secondary Outcome: Sensory Organization Test (SOT) Vestibular
Description: The SOT assesses the sensory components of balance by measuring postural sway balance in different conditions as a useful predictor of fall risk. The ratio score indicates ability to maintain balance in the presence of inaccurate visual cues. Scores are represented as a percentage from 0 to 100, with scores closer to 100 indicating greater stability.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent stability maintained
Arm/Group | Health Education | Yoga
Number analyzed (Participants) | 21 | 20
percent stability maintained | -1.1 (23.8) | 8.9 (29.1)

5. Secondary Outcome: Limits of Stability (LOS)
Description: The LOS is used to define a participant's "cone of stability" and measures components of balance and stability related to reaction time, directional control, and the ability to make corrective movements. Movement velocity indicates the speed of center of gravity (COG) displacement in degrees per second, with higher values signifying quicker movement through the region of stability.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | Health Education | Yoga
Number analyzed (Participants) | 21 | 20
degrees per second | -0.62 (1.62) | 0.51 (1.61)

6. Secondary Outcome: Grip Strength
Description: Grip Strength was assessed with an adjustable, hydraulic grip strength dynamometer.(26) The measure uses the average of two trials for both the left and right hand.
Time Frame: Change from baseline to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pounds of pressure
Arm/Group | Yoga | Health Education
Number analyzed (Participants) | 20 | 21
pounds of pressure | 0.12 (8.03) | -5.2 (11.72)

7. Secondary Outcome: SF-36
Description: The SF-36 has 36 items and takes about 8-10 minutes to complete. The scale measure domains of health-related quality of life and two summary scores corresponding to physical and mental health. Scores for each subscale are standardized and range from 0-100 with higher scores representing better quality of life.
Time Frame: Change from baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Health Education
Number analyzed (Participants) | 22 | 23
units on a scale
  Physical | 0.23 (5.99) | -1.2 (5.21)
  Mental | 0.7 (5.6) | -3.2 (7.7)

8. Secondary Outcome: Center for Epidemiologic Studies Short Depression Scale (CES-D 10)
Description: Depression was assessed using the 10-item Center for Epidemiologic Studies Short Depression Scale (CES-D 10). Scores can range from 0-30 with higher scores indicating higher levels of depressive symptoms.
Time Frame: Change from baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Health Education
Number analyzed (Participants) | 22 | 23
units on a scale | -0.35 (3.15) | 1.14 (3.59)

9. Secondary Outcome: Brief Anxiety Inventory (BAI)
Description: Anxiety was assessed using the Brief Anxiety Inventory (BAI). The self-administered BAI consists of 21 items, and has well-established reliability(29) and validity. Scores can range from 0-63 with higher scores indicating greater levels of anxiety.
Time Frame: Change from baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Health Education
Number analyzed (Participants) | 22 | 23
units on a scale | 0.18 (7.48) | 2.87 (5.89)

10. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Sleep quality was measured using the Pittsburgh Sleep Quality Index (PSQI). The measure has 21 items and scores can range from 0-21 with higher scores indicating lower sleep quality.
Time Frame: Change from baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga | Health Education
Number analyzed (Participants) | 22 | 23
units on a scale | -0.5 (2.52) | -0.2 (2.27)

11. Secondary Outcome: Participant Satisfaction
Description: Participant Satisfaction with participation was rated on a 0-10 scale (10 = most positive) usingquestions about enjoyment with and benefits of participation.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Education | Yoga
Number analyzed (Participants) | 23 | 22
units on a scale | 8.1 (2.7) | 8.4 (2.8)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Yoga | Health Education
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 13/22 | 9/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga (N=22) | Health Education (N=24)
Increased pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes